CLINICAL TRIAL: NCT05500807
Title: Emicizumab for Severe VON Willebrand Disease (VWD) and VWD/Hemophilia A
Acronym: BCDI-XII
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bleeding and Clotting Disorders Institute Peoria, Illinois (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jonathan Roberts, Associate Medical Director, Bleeding and Clotting Disorders Institute Peoria, Illinois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCDI-XII
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2024-12

CONDITIONS: Von Willebrand Disease, Type 3; Concomitant VWD and Hemophilia
MeSH Terms: conditions — von Willebrand Disease, Type 3; Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Intervention Model Description: 40 patients who will receive emicizumab prophylactically
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label Emicizumab (Other): Emicizumab prophylaxis
  Interventions: Drug: Emicizumab

INTERVENTIONS:
Drug: Emicizumab — Subcutaneous injection of emicizumab for prophylaxis
  Other Names: Hemlibra

SUMMARY:
Von Willebrand Disease (VWD) is the most common inherited bleeding disorder affecting up to 0.1% of the population, is usually characterized by mucocutaneous bleeding, HMB, surgical bleeding or other hemostatic challenges. Severe bleeding events require VWF concentrates administered solely through intravenous access. Emicizumab (Hemlibra) is a monoclonal bispecific antibody developed to bind activated FIX and FX and mimic FVIII cofactor functionality. Hemlibra is administered via subcutaneous injection rather than intravenous infusion. The hypothesis of this study is that Emicizumab is safe and efficacious for prophylaxis in severe VWD and concomitant VWD/hemophilia patients.

DETAILED DESCRIPTION:
Von Willebrand Disease (VWD) is the most common inherited bleeding disorder affecting up to 0.1% of the population, is usually characterized by mucocutaneous bleeding, HMB, surgical bleeding or other hemostatic challenges. VWD currently has few therapies generally useful in management of bleeding events including antifibrinolytics, desmopressin (DDAVP), and VWF concentrates, which may be plasma-derived (VWF with and without FVIII) or recombinant. Minor bleeding may be successfully treated with antifibrinolytics and DDAVP; however, more severe bleeding requires VWF concentrates that are administered solely through intravenous access.

Similarly, it can be challenging to treat concomitant bleeding disorders with the existing therapeutic options available, and patients with concurrent VWD and hemophilia A primarily have VWF/FVIII concentrate or desmopressin (DDAVP) available for treatment. It has been well-recognized that patients, caregivers, and medical providers desire additional, simplified therapeutic options that are not intravenous to treat severe bleeding disorders. Therefore, a simplified, subcutaneous therapeutic that prevents bleeding would be strongly desired. Though its use in the hemophilia A population is growing, additional potential emicizumab applications for hemostatic control in other hemostatic disorders remain unknown. A recent case report highlighted the hemostatic efficacy of emicizumab off-label use in type 3 von Willebrand Disease (VWD), another severe bleeding disorder. This pediatric patient had type 3 VWD with alloantibodies and a bleeding phenotype similar to hemophilia A with inhibitor patients, requiring suboptimal bleeding management with rFVIIa and activated prothrombin complex concentrates (aPCC). Emicizumab prophylaxis was initiated and the patient no longer required aPCC prophylaxis and rare use of rFVIIa for acute bleeding events (only 1 trauma-induced soft tissue hematoma at the time of publication). The authors concluded their report suggested the bleeding phenotype in type 3 VWD is expressed mainly due to factor VIII deficiency. This study suggests a potential additional application for emicizumab in severe VWD.

A pilot multicenter, prospective open-label study of emicizumab prophylaxis in severe VWD and concomitant VWD/hemophilia A. Patients will have a one-year retrospective chart review of annualized bleed rate and hemostatic therapies collected at the time of enrollment. Patients will then be treated with emicizumab with 3mg/kg weekly for 4 weeks loading dose, followed by once weekly prophylaxis of 1.5mg/kg for 1 year. Per emicizumab FDA-approved prescribing information for hemophilia A, dose up-titration to 3 mg/kg once weekly will be allowed after 24 weeks on HEMLIBRA prophylaxis in case of suboptimal efficacy (i.e., ≥ 2 spontaneous and clinically significant bleeds) Treatment records will be maintained along with bleeding event logs. Breakthrough bleeding events may be treated with the patients usual on-demand therapy with antifibrinolytics or VWF/FVIII concentrates per clinician discretion. Patient reported outcome assessments will be collected throughout the clinical study to collect impact of the treatment on the individual patients, assessing quality of life, physical, emotional, social and general symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 0 and older (infants weighing ≥3 kg)
* ability to comply with protocol in investigators judgement
* diagnosis of: severe VWD type 3, or VWD with VWF antigen, activity or collagen binding </= 20 U/dl or variant VWD confirmed by genetic mutation and VWF ag, activity or CB < 50 U/dl based on historical medical records of study site.
* diagnosis of VWD/hemophilia A defined as VWF:ag, activity or CB <50 U/dl, and mild moderate or severe hemophilia A(defined by ISTH criteria) based on historical medical records of the study site.
* plan to be adherent to emicizumab prophylaxis during the study
* Patient's bleeding phenotype necessitating prophylaxis per treating provider recommendations.
* Patient on current prophylaxis for VWD or VWD/hemophilia A may enroll if they are currently on a non-emicizumab agent, and if it has been > 18 months since last off-label dose of emicizumab, and are willing to discontinue current prophylaxis.
* For menstruating individuals: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the study period. A menstruating individual is considered to be of childbearing potential if they are post-menarchal, have not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and have not undergone surgical sterilization (removal of ovaries and/or uterus).

Examples of highly effective contraceptive methods with a failure rate of < 1% per year include proper use of combined oral or injected hormonal contraceptive, bilateral tubal ligation, male sterilization, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Patients and/or infants weighing < 3 kg.
* Patients with low VWF or non-severe VWD (ie.not meeting the above criteria)
* Other concomitant bleeding disorders including coagulopathy from liver cirrhosis.
* Current treatment with emicizumab or emicizumab therapy in the previous 18 months.
* Previous (in the past 12 months) or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or current signs of thromboembolic disease
* Other conditions (e.g., certain autoimmune diseases, including, but not limited to diseases such as systemic lupus erythematosus, inflammatory bowel disease, and antiphospholipid syndrome) that may increase the risk of bleeding or thrombosis
* Patients who are at high risk for thrombotic microangiopathy (TMA; e.g., have a previous medical or family history of TMA), in the investigator's judgment
* Would refuse treatment with blood or blood products, if necessary.
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study
* Treatment with any of the following:

An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration before Study Day 1 A non-hemophilia-related investigational drug within the last 30 days or 5 halflives- before Study Day 1, whichever is longer An investigational drug concurrently

* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection
* Pregnant or lactating, or intending to become pregnant during the study
* Women of childbearing potential must have a negative serum pregnancy test result within 7 days before Study Day 1
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Serious infection requiring oral or IV antibiotics within 30 days prior to screening

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Emicizumab is efficacious for prophylaxis in severe VWD & concomitant VWD/hemophilia A | 18 months
  Establish bleed occurrence during treatment evaluated through descriptive statistical analysis to determine proof of principle
Emicizumab is safe for prophylaxis in severe VWD & concomitant VWD/Hemophilia A | 18 months
  Collection of AE's, hypersensitivity reactions, thrombotic events during treatment

SECONDARY OUTCOMES:
Reduced treatment burden vs VWF/FVIII prophylaxis | 18 months
  # of infusions and methods of infusions collected during study
Decreased bleed occurrence | 12 months
  Evaluate historical ABR with on demand or prophy prior to study treatment
Diminish bleed severity | 18 months
  Collection of bleed data prior to study entry and throughout study treatment

OTHER OUTCOMES:
Improve health related QOL in study participants | 18 months
  Collection of HRQOL PRO's
Reduce product use for spontaneous or traumatic bleeds | 18 months
  Bleed & treatment logs collecting product use prior to study entry and throughout study treatment
Reduce product use during surgery | 18 months
  Bleed & treatment logs collect information for any surgical procedure while on study, blood loss, hemostatic efficacy and concentrate consumption.
Reduce self-reported treatment burden for HMB | 18 months
  Bleed & treatment logs collect treatment information prior to and during study for HMB including antifibrinolytics, concentrates and hormonal therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan C Roberts, MD, Principal Investigator — Bleeding and Clotting Disorders Institute
Locations (9):
- United States (9):
  - The Center for Comprehensive Care and Diagnosis of Inherited Blood Disorders (CIBD), Orange, California
  - Stanford University: Stanford Children's Health, Redwood City, California
  - University of Miami - Miller School of Medicine, Coral Gables, Florida
  - St. Joseph's Children's Hospital - Center for Bleeding and Clotting Disorders, Tampa, Florida
  - Bleeding and Clotting Disorders Institute (BCDI), Peoria, Illinois
  - Innovative Hematology, Inc. (IHI), Indianapolis, Indiana
  - University of Michigan Medical School, Ann Arbor, Michigan
  - Central Michigan University: Children's Hospital of Michigan, Mount Pleasant, Michigan
  - Washington Center for Bleeding Disorders, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Handorf CR. Background--setting the stage for alternate-site laboratory testing. Clin Lab Med. 1994 Sep;14(3):451-8. PMID 7805340
- [Background] Kaminaga T, Nishimura T, Hayashida K, Ishida Y, Hiroki M. Clinical application of spontaneous red blood cell labeling with Tc-99m sodium pertechnetate. Clin Nucl Med. 1994 Oct;19(10):895-7. doi: 10.1097/00003072-199410000-00012. PMID 7805326
- [Background] Rodeghiero F, Castaman G, Dini E. Epidemiological investigation of the prevalence of von Willebrand's disease. Blood. 1987 Feb;69(2):454-9. PMID 3492222
- [Background] Werner EJ, Broxson EH, Tucker EL, Giroux DS, Shults J, Abshire TC. Prevalence of von Willebrand disease in children: a multiethnic study. J Pediatr. 1993 Dec;123(6):893-8. doi: 10.1016/s0022-3476(05)80384-1. PMID 8229521
- [Background] Shima K. [Endless voyage. The life of Ms. Shin Tanaka. 6. Chapter 2]. Josanpu Zasshi. 1982 Dec;36(12):1036-43. No abstract available. Japanese. PMID 6759735
- [Background] Roberts JC, Morateck PA, Christopherson PA, Yan K, Hoffmann RG, Gill JC, Montgomery RR; Zimmerman Program Investigators. Rapid discrimination of the phenotypic variants of von Willebrand disease. Blood. 2016 May 19;127(20):2472-80. doi: 10.1182/blood-2015-11-664680. Epub 2016 Feb 25. PMID 26917779
- [Background] Miller CH, Hilgartner MW, Harris MB, Bussel JB, Aledort LM. Concurrence of von Willebrand's disease and hemophilia A: implications for carrier detection and prevalence. Am J Med Genet. 1986 May;24(1):83-94. doi: 10.1002/ajmg.1320240110. PMID 3085499
- [Background] Casonato A, Pontara E, Boscaro M, Dannhauser D, Sartori MT, Girolami A. Combined haemophilia A and type I von Willebrand's disease: a family study including an evaluation of the effects of DDAVP infusion. Haematologia (Budap). 1993;25(1):57-67. PMID 8339998
- [Background] Kitazawa T, Igawa T, Sampei Z, Muto A, Kojima T, Soeda T, Yoshihashi K, Okuyama-Nishida Y, Saito H, Tsunoda H, Suzuki T, Adachi H, Miyazaki T, Ishii S, Kamata-Sakurai M, Iida T, Harada A, Esaki K, Funaki M, Moriyama C, Tanaka E, Kikuchi Y, Wakabayashi T, Wada M, Goto M, Toyoda T, Ueyama A, Suzuki S, Haraya K, Tachibana T, Kawabe Y, Shima M, Yoshioka A, Hattori K. A bispecific antibody to factors IXa and X restores factor VIII hemostatic activity in a hemophilia A model. Nat Med. 2012 Oct;18(10):1570-4. doi: 10.1038/nm.2942. Epub 2012 Sep 30. PMID 23023498
- [Background] Shima M, Hanabusa H, Taki M, Matsushita T, Sato T, Fukutake K, Fukazawa N, Yoneyama K, Yoshida H, Nogami K. Factor VIII-Mimetic Function of Humanized Bispecific Antibody in Hemophilia A. N Engl J Med. 2016 May 26;374(21):2044-53. doi: 10.1056/NEJMoa1511769. PMID 27223146
- [Background] Uchida N, Sambe T, Yoneyama K, Fukazawa N, Kawanishi T, Kobayashi S, Shima M. A first-in-human phase 1 study of ACE910, a novel factor VIII-mimetic bispecific antibody, in healthy subjects. Blood. 2016 Mar 31;127(13):1633-41. doi: 10.1182/blood-2015-06-650226. Epub 2015 Dec 1. PMID 26626991
- [Background] Oldenburg J, Mahlangu JN, Kim B, Schmitt C, Callaghan MU, Young G, Santagostino E, Kruse-Jarres R, Negrier C, Kessler C, Valente N, Asikanius E, Levy GG, Windyga J, Shima M. Emicizumab Prophylaxis in Hemophilia A with Inhibitors. N Engl J Med. 2017 Aug 31;377(9):809-818. doi: 10.1056/NEJMoa1703068. Epub 2017 Jul 10. PMID 28691557
- [Background] Mahlangu J, Oldenburg J, Paz-Priel I, Negrier C, Niggli M, Mancuso ME, Schmitt C, Jimenez-Yuste V, Kempton C, Dhalluin C, Callaghan MU, Bujan W, Shima M, Adamkewicz JI, Asikanius E, Levy GG, Kruse-Jarres R. Emicizumab Prophylaxis in Patients Who Have Hemophilia A without Inhibitors. N Engl J Med. 2018 Aug 30;379(9):811-822. doi: 10.1056/NEJMoa1803550. PMID 30157389
- [Background] Levy GG, Asikanius E, Kuebler P, Benchikh El Fegoun S, Esbjerg S, Seremetis S. Safety analysis of rFVIIa with emicizumab dosing in congenital hemophilia A with inhibitors: Experience from the HAVEN clinical program. J Thromb Haemost. 2019 Sep;17(9):1470-1477. doi: 10.1111/jth.14491. Epub 2019 Jun 17. PMID 31124272
- [Background] Petrini P. Identifying and overcoming barriers to prophylaxis in the management of haemophilia. Haemophilia. 2007 Sep;13 Suppl 2:16-22. doi: 10.1111/j.1365-2516.2007.01501.x. PMID 17685919
- [Background] Saccullo G, Makris M. Prophylaxis in von Willebrand Disease: Coming of Age? Semin Thromb Hemost. 2016 Jul;42(5):498-506. doi: 10.1055/s-0036-1581106. Epub 2016 Jun 2. PMID 27253087
- [Background] Berntorp E. Prophylaxis in von Willebrand disease. Haemophilia. 2008 Nov;14 Suppl 5:47-53. doi: 10.1111/j.1365-2516.2008.01851.x. PMID 18786010
- [Background] Federici AB. Prophylaxis in patients with von Willebrand disease: who, when, how? J Thromb Haemost. 2015 Sep;13(9):1581-4. doi: 10.1111/jth.13036. Epub 2015 Jul 28. No abstract available. PMID 26081061
- [Background] Makris M, Oldenburg J, Mauser-Bunschoten EP, Peerlinck K, Castaman G, Fijnvandraat K; subcommittee on Factor VIII, Factor IX and Rare Bleeding Disorders. The definition, diagnosis and management of mild hemophilia A: communication from the SSC of the ISTH. J Thromb Haemost. 2018 Dec;16(12):2530-2533. doi: 10.1111/jth.14315. Epub 2018 Nov 15. No abstract available. PMID 30430726